CLINICAL TRIAL: NCT05873335
Title: In Vivo Testing for SpO2 Accuracy on Healthy Adults Under Laboratory Conditions
Brief Title: In Vivo Pulse Oximeter Validation Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gabi SmartCare (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: SpO2_3
Record Dates: First submitted 2023-05-04; First posted 2023-05-24 (Actual); Results first posted 2024-12-12 (Actual); Last update posted 2024-12-12 (Actual); Status verified 2024-12

CONDITIONS: Hypoxia
MeSH Terms: conditions — Hypoxia | interventions — Air; Carbon Dioxide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Healthy Adults (Experimental): Healthy adults
  Interventions: Combination Product: Mixtures of nitrogen, air, and carbon dioxide

INTERVENTIONS:
Combination Product: Mixtures of nitrogen, air, and carbon dioxide — Hypoxia was induced to different and stable levels of oxyhemoglobin saturation (between 70-100%) by having subjects breathe mixtures of nitrogen, air, and carbon dioxide controlled by the study physician by adjusting gas flows with valves according to breath-by-breath estimates of oxygen saturation calculated from end-tidal PO2 and PCO2 displayed on a screen using LabVIEW 2015
  Other Names: Radial arterial cannula

SUMMARY:
The goal of this clinical trial is to compare values of SpO2 provided by the DUT and the SaO2 used as a reference in healthy adults. The main question it aims to answer is: what is the accuracy of the subject device compared to the 510(k)-cleared reference device

A radial arterial cannula was placed in the wrist of each subject for arterial blood sampling and a subject device was placed on each arm of the patients. Then, hypoxia was induced to different stable levels of oxyhemoglobin saturation between 70-100% by having subjects breathe mixtures of nitrogen, air, and carbon dioxide controlled by the study physician. Values of SpO2 and SaO2 were then compared to provide a root mean square error and conclude on the subject device accuracy.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult
* Normal hemoglobin levels (Hemoglobin > 10 g/dL)

Exclusion Criteria:

* Systemic illness
* Obesity

Ages: 21 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2023-02-28 (Actual); Primary Completion 2023-03-01 (Actual); Study Completion 2023-03-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Philip E Bickler, M.D., PhD., Principal Investigator — University of California, San Francisco
Locations (1):
- Hypoxia Research Laboratory, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Healthy Adults: Healthy adults
  Mixtures of nitrogen, air, and carbon dioxide: Hypoxia was induced to different and stable levels of oxyhemoglobin saturation (between 70-100%) by having subjects breathe mixtures of nitrogen, air, and carbon dioxide controlled by the study physician by adjusting gas flows with valves according to breath-by-breath estimates of oxygen saturation calculated from end-tidal PO2 and PCO2 displayed on a screen using LabVIEW 2015. 2 Gabi Band devices were placed on the subject (one on each arm). It was expected that the Accuracy Root Mean Square (ARMS) performance of the oximetry system would meet the required specification of ARMS of 3.5% or less.
Period: Overall Study
Arm/Group | Healthy Adults
Started | 12
Completed | 12
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: 12 healthy adults in total, each wearing 1 Gabi Band device on each arm
Arm/Group | Healthy Adults
Number analyzed (Participants) | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 12
  >=65 years | 0
Age, Continuous [Mean (Full Range); unit: years] | 25.25 [22 to 28]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 5
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 3
  More than one race | 1
  Unknown or Not Reported | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 12

OUTCOME MEASURES:

1. Primary Outcome: Measure of Accuracy (ARMS [%])
Description: Arms, given in percentage or rms error, is the calculation of root mean square between SpO2 values from the subject device and the SaO2 from the Hemoximeter. It is a way of averaging the absolute values of errors over the full measurement range and is a similar measurmeent to a "rms error". It indicates how far (accurate) the provided value is from the reference used.
Time Frame: 1 hour
Measure: Number; unit: Percentage
Arm/Group | Healthy Adults
Number analyzed (Participants) | 12
Percentage | 2.95

ADVERSE EVENTS:
Time Frame: 2 hours
Description: All healthy participants
Arm/Group | Healthy Adults
All-Cause Mortality (participants affected / at risk) | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12
Other Adverse Events (participants affected / at risk) | 0/12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-02-02): https://cdn.clinicaltrials.gov/large-docs/35/NCT05873335/Prot_SAP_002.pdf